CLINICAL TRIAL: NCT07359313
Title: Incidence of Colon Ischemia in Patients After Cardiopulmonary Resuscitation (CPR): a Prospective Single-center Epidemiological Incidence Study
Brief Title: Incidence of Colon Ischemia in Patients After Cardiopulmonary Resuscitation (CPR)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, PD Dr. Alexander Supady, Senior Physician, University Hospital Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-1320-S1
Record Dates: First submitted 2025-12-19; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest (CA)
Keywords: cardiac arrest; cardiopulmonary resuscitation; CPR; extracorporeal cardiopulmonary resuscitation; ECPR; VA ECMO; colonoscopy; mesenteric ischemia
MeSH Terms: conditions — Heart Arrest; Mesenteric Ischemia | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: Prospective epidemiological incidence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- early colonoscopy after successful CPR (Other): bedside colonoscopy 24-36 hours after successful CPR
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — bedside colonoscopy without bowel cleansing early (24-36h) after successful CPR

SUMMARY:
Bedside colonoscopy 24-36 hours after successful CPR

DETAILED DESCRIPTION:
According to previous observations, many patients after CPR develop acute non-occlusive mesenteric ischemia. However, due to the lack of established screening strategies, the number of unreported cases may be high. Routine colonoscopy at 24-36 hours after CPR may be a safe, easy and cost-effective strategy for early detection of severe mesenteric ischemia and transfer to surgical treatment. However, this strategy has not been formally evaluated in larger prospective cohorts. In our center, we perform routine colonoscopy at 24 to 36 hours after cardiac arrest in all patients who receive extracorporeal CPR (ECPR), i.e., in all patients with prolonged cardiac arrest refractory to conventional CPR measures who therefore receive venoarterial extracorporeal membrane oxygenation (VA ECMO) for cardiocirculatory support. In these patients, colonoscopy screening was feasible and safe, and our data suggest clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 18 years) admitted to the participating department AND
* in-hospital or out-of-hospital cardiac arrest (IHCA, OHCA)

Exclusion Criteria:

* resuscitation period of ≤ 5 minutes
* awake and contactable patients (GCS ≥ 13)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2028-01-06 (Estimated); Study Completion 2028-02-06 (Estimated)

PRIMARY OUTCOMES:
Detection of colon ischemia | from baseline (0 hours) until day 30
  Detection of colon ischemia within 30 days after return of spontaneous circulation

SECONDARY OUTCOMES:
in-hospital mortality | from baseline (0 hours) until hospital discharge
  in-hospital mortality
abdominal surgery ((hemi-)colectomy) | from baseline (0 hours) until hospital discharge
  number of patients requiring/receiving abdominal surgery ((hemi-)colectomy)
functional outcome | day 30, day 60 and day 90
  Cerebral Performance Category (CPC)
Liver function | within 0-72 hours after CPR
  Liver function parameters: Quick/INR, AST, ALT, AP, g-GT
renal function | within 0-72 hours after CPR
  Renal function parameters: creatinine, BUN
Urine output | within 0-72 hours after CPR
  Urine output (ml)
Renal replacement therapy | from baseline (day 0) until day 30
  Implementation of renal replacement therapy within 30 days after return of spontaneous circulation
Serum lactate | within 0-72 hours after CPR
  Serum lactate
SOFA score | at 0 hours, 24 hours, 48 hours, 72 hours after CPR
  SOFA
SAPS II score | at 0 hours, 24 hours, 48 hours, 72 hours after CPR
  SAPS II

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center - University of Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No